CLINICAL TRIAL: NCT00046319
Title: A Phase II, Randomized, Double-Blind, Dose-Controlled, Dose-Ranging, Multicenter Study of BSF 208075 Evaluating Exercise Capacity in Patients With Moderate to Severe Pulmonary Arterial Hypertension
Brief Title: Study of BSF 208075 Evaluating Exercise Capacity in Patients With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMB-220
Record Dates: First submitted 2002-09-26; First posted 2002-09-30 (Estimated); Last update posted 2009-04-16 (Estimated); Status verified 2009-04

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension; Primary Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension | interventions — ambrisentan

INTERVENTIONS:
Drug: BSF 208075

SUMMARY:
The purpose of this study is to determine if treating patients suffering from moderate to severe pulmonary arterial hypertension with BSF 208075 will improve the patients' ability to exercise.

DETAILED DESCRIPTION:
This is a randomized, double-blind study evaluating the effectiveness of BSF 208075 in treating patients with moderate to severe pulmonary hypertension. A four-week Screening Period will be followed by 12 weeks of Treatment. After a subject qualifies for the study, the subject will be randomized to one of four doses of BSF 208075 (1.0, 2.5, 5.0 or 10.0 mg po qd). Subjects randomized to the 1.0 or 2.5 mg dose groups will receive their respective doses of BSF 208075 each day throughout the 12-week Treatment Period. Subjects in the two other dose groups will begin treatment at 2.5 mg per day for two weeks and then their dose will be increased to 5.0 mg for an additional two weeks. After two weeks of treatment at 5.0 mg, subjects randomized to the 10.0 mg dose group will undergo a final up-titration. After reaching the randomized dose level, subjects will receive their assigned dose throughout the Treatment Period. Subjects will remain on the randomized treatment through Week 12. In the event that a subject is not tolerating study drug, dose adjustment is permitted during the Treatment Period. Upon completion of the 12-week Treatment Period subjects will either complete a four-week Down-titration Period or enter an optional 12-week Open-label Extension. All subjects that choose to participate in the Open-label Extension will be unblinded and have their dose of BSF 208075 optimized based on the subjects response during the Treatment Period.

ELIGIBILITY:
--Disease Characteristics--

* Current diagnosis of either PPH or PAH secondary to the scleroderma spectrum of disease (e.g., mixed connective tissue disease, systemic lupus erythematosus, systemic sclerosis, or overlap syndrome), anorexigen use, or human immunodeficiency virus (HIV) infection at the time of screening
* By means of a right heart catheterization, completed prior to Screening Visit subjects must meet all of the following hemodynamic criteria:

  * Mean pulmonary arterial pressure of >/= 25 mmHg
  * Pulmonary vascular resistance >3 mmHg/L/min
  * Pulmonary capillary wedge pressure or left ventricle end diastolic pressure of <15 mmHg
* Stable on conventional therapy for PAH, including diuretics, digoxin, or supplemental oxygen, for at least one month prior to the Screening Visit
* Subjects with a diagnosis of HIV must have stable disease status at the time of screening. The subject may be enrolled if they meet the definition of a stable HIV status defined as:

  * No addition of medications for treatment of HIV in the last two months
  * No active opportunistic infection at the time of screening
  * No hospitalizations due to HIV within the past four weeks
* Able to walk at least 150 meters, but no more than 450 meters, in a six minute walk test at the time of the Screening Visit
* No pulmonary arterial hypertension due to or associated with congenital heart disease, interstitial lung disease, chronic obstructive pulmonary disease, or chronic thrombotic and/or embolic disease, as documented by a historical echocardiogram, chest X-ray, ventilation/perfusion (V/Q) scan, and/or pulmonary arteriogram
* No subjects who have, as measured by a historical pulmonary function test:

  * Total lung capacity (TLC) <70% of predicted normal or;
  * Forced expiratory volume in one second (FEV1) <65% of predicted normal

--Other Criteria--

* Subjects are excluded if they have:

  * A serum ALT or AST lab value that is greater than 1.5 times the upper limit of normal at any time during the Screening Period
  * Contraindication to treatment with an endothelin receptor antagonist
  * Demonstrated noncompliance with previous medical regimens
  * A recent history of abusing alcohol or illicit drugs
  * Participated in a clinical study involving another investigational drug or device within four weeks before the Screening Visit or at any time during the study

--Patient Characteristics--

* Women of childbearing potential must:

  * Have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at the Randomization Visit. Women who are surgically sterile or those who are post-menopausal for at least two years are not considered to be of childbearing potential
  * Agree to use a reliable double barrier method of contraception until study completion and for at least four weeks following their final study visit
* All males must be informed of the potential risks of testicular tubular atrophy and infertility associated with taking this study drug and queried regarding his understanding of the potential risks as described in the Informed Consent Form

Excluded:

* Pregnant or breastfeeding
* Have a history of malignancies within the past five years, with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix
* Any other disease which, in the investigators opinion, may adversely affect the safety of the subject and/or efficacy of the study drug or severely limit the lifespan of the subject

--Prior/Concurrent Therapy--

* Stable on conventional therapy for PAH, including diuretics, digoxin, or supplemental oxygen, for at least one month prior to the Screening Visit

Excluded Therapies:

* IV inotropes within two weeks prior to the Screening Visit
* Chronic prostanoid therapy (epoprostenol, treprostinil, iloprost, beraprost, or any other investigational prostacyclin derivative) within four weeks prior to the Screening Visit
* Bosentan within four weeks prior to the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-09; Study Completion 2003-06

PRIMARY OUTCOMES:
Change from baseline to Week 12 in six minute walk distance

SECONDARY OUTCOMES:
Change from baseline to Week 12 in:
Borg Dyspnea Index
WHO Functional Classification
Subject Global Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Rubin, MD, Principal Investigator — UCSD Medical Center
Locations (21):
- United States (15):
  - University of Southern California, Los Angeles, California
  - University of California San Diego Medical Center, San Diego, California
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Los Angeles County Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Rush Presbyterian, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian Hospital, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Heart Care Associates, Milwaukee, Wisconsin
- St. Vincent's Hospital, Sydney, Australia
- Erasmus University, Brussels, Belgium
- Hopital Antoine Beclere, Clamart, Cedex, France
- Germany (2):
  - University of Giessen, Giessen
  - Hannover Medical School, Hanover
- University of Bologna - Institute of Cardiology, Bologna, Italy